CLINICAL TRIAL: NCT05432115
Title: Bismuth Quadruple Therapy for Helicobacter Pylori Rescue Therapy: A Multicenter Randomized Non-Inferiority Trial of Different Tetracycline Doses and Frequencies.
Brief Title: Bismuth Quadruple Therapy for Helicobacter Pylori Rescue Therapy of Different Tetracycline Doses and Frequencies.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Collaborators: Peking University Care Luzhong Hospital (Other); Zibo Central Hospital (Other Government); Zhengzhou Central Hospital (Other); Taierzhuang District People's Hospital (Other); Yuncheng Traditional Chinese Medicine Hospital (Other)
Responsible Party: Principal Investigator, Yanqing Li, Dr, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022032
Record Dates: First submitted 2022-06-20; First posted 2022-06-27 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; tetracycline; bismuth quadruple therapy
MeSH Terms: interventions — Tetracycline; Amoxicillin; Esomeprazole; Bismuth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tid group (Experimental): Tid group: Amoxicillin 1000mg bid+ Tetracycline 500mg tid+ Bismuth + Esomeprazole 40mg bid
  Interventions: Drug: Tetracyclin
- Qid group (Active Comparator): Qid group: Amoxicillin 1000mg bid+ Tetracycline 500mg qid+ Bismuth + Esomeprazole 40mg bid
  Interventions: Drug: Tetracyclin

INTERVENTIONS:
Drug: Tetracyclin — Amoxicillin 1000mg bid +Tetracycline 500mg tid/qid +Bismuth+Esomeprazole 40mg bid
  Other Names: Amoxicillin; Esomeprazole; Bismuth

SUMMARY:
The researchers collect H.pylori-positive patients who need rescue therapy from the outpatient clinic. The subjects were randomized to receive a dose and frequency of tetracycline 500mg tid or qid of bismuth quadruple eradication therapy. 6-8 weeks after treatment, the subjects will re-take the 13C-urea breath test. Calculate the eradication rates, adverse reaction rates and patient compliance of each group.

DETAILED DESCRIPTION:
The researchers collect H.pylori-positive patients who need rescue therapy from the outpatient clinic. If the subject meets the selection criteria but not the exclusion criteria, and signs an informed consent form, the researchers randomized the subjects in groups: subjects received a dose and frequency of tetracycline 500mg tid or qid of bismuth quadruple eradication therapy. The medication of groups are as follows. 6-8 weeks after the eradication treatment, the subjects will review the 13C-urea breath test, and the researcher records the results.

After all subjects were tested, the eradication rates, adverse reaction rates and patient compliance of each group were calculated.

According to the dose and frequency of tetracycline, it is randomized into a tid treatment group and a qid treatment group. The two groups of bismuth quadruple regimens are the same, as follows:

Tid group: Amoxicillin 1000mg bid+ Tetracycline 500mg tid+ Bismuth + Esomeprazole 40mg bid Qid group: Amoxicillin 1000mg bid+ Tetracycline 500mg qid+ Bismuth + Esomeprazole 40mg bid

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-70.
2. Patients with H.pylori infection (Positive for rapid urease test or 13C/14C-urea breath test).
3. Patients who have previous failed H. pylori eradication treatment, and ≤ 2 times.

Exclusion Criteria:

1. Patients with serious underlying diseases, such as liver insufficiency (Aspartate aminotransferase or alanine aminotransferase greater than 1.5 times the normal value), renal insufficiency (Cr≥2.0mg/dL or glomerular filtration rate <50 ml/min), immunosuppression, malignant tumors, Coronary heart disease or coronary artery stenosis ≥75%.
2. Patients who are pregnant or lactating or unwilling to take contraceptive measures during the trial.
3. Patients with active gastrointestinal bleeding.
4. Patients with a history of upper gastrointestinal surgery.
5. Patients allergic to treatment drugs.
6. Patients with medication history of bismuth agents, antibiotics, proton pump inhibitor and other drugs within 4 weeks
7. Patients with other behaviors that may increase the risk of illness, such as alcohol and drug abuse
8. Patients who are unwilling or incapable to provide informed consents

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Estimated)
Dates: Start 2022-06-25 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Eradication rate | Immediately after follow-up check
  Both intention to treat (ITT) and per-protocol (PP) analyses will be used for the assessment of the eradication rates of Helicobacter pylori infections in two groups. The ITT analysis includes all randomly assigned patients who take at least one dose of the study medications. The PP analysis is limited to patients who take over 90% of the study medications and complete follow-up.

SECONDARY OUTCOMES:
Rate of adverse reactions | Immediately after follow-up check
  Rate of adverse reactions
Patient compliance | Immediately after follow-up check
  Good compliance is defined as the actual dosage is within the range of 80%-100% of the dosage that should be taken.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital, Jinan, Shandong, China

REFERENCES:
- [Result] Hooi JKY, Lai WY, Ng WK, Suen MMY, Underwood FE, Tanyingoh D, Malfertheiner P, Graham DY, Wong VWS, Wu JCY, Chan FKL, Sung JJY, Kaplan GG, Ng SC. Global Prevalence of Helicobacter pylori Infection: Systematic Review and Meta-Analysis. Gastroenterology. 2017 Aug;153(2):420-429. doi: 10.1053/j.gastro.2017.04.022. Epub 2017 Apr 27. PMID 28456631
- [Result] Malfertheiner P, Megraud F, O'Morain CA, Gisbert JP, Kuipers EJ, Axon AT, Bazzoli F, Gasbarrini A, Atherton J, Graham DY, Hunt R, Moayyedi P, Rokkas T, Rugge M, Selgrad M, Suerbaum S, Sugano K, El-Omar EM; European Helicobacter and Microbiota Study Group and Consensus panel. Management of Helicobacter pylori infection-the Maastricht V/Florence Consensus Report. Gut. 2017 Jan;66(1):6-30. doi: 10.1136/gutjnl-2016-312288. Epub 2016 Oct 5. PMID 27707777
- [Result] Ding SZ, Du YQ, Lu H, Wang WH, Cheng H, Chen SY, Chen MH, Chen WC, Chen Y, Fang JY, Gao HJ, Guo MZ, Han Y, Hou XH, Hu FL, Jiang B, Jiang HX, Lan CH, Li JN, Li Y, Li YQ, Liu J, Li YM, Lyu B, Lu YY, Miao YL, Nie YZ, Qian JM, Sheng JQ, Tang CW, Wang F, Wang HH, Wang JB, Wang JT, Wang JP, Wang XH, Wu KC, Xia XZ, Xie WF, Xie Y, Xu JM, Yang CQ, Yang GB, Yuan Y, Zeng ZR, Zhang BY, Zhang GY, Zhang GX, Zhang JZ, Zhang ZY, Zheng PY, Zhu Y, Zuo XL, Zhou LY, Lyu NH, Yang YS, Li ZS; National Clinical Research Center for Digestive Diseases (Shanghai), Gastrointestinal Early Cancer Prevention & Treatment Alliance of China (GECA), Helicobacter pylori Study Group of Chinese Society of Gastroenterology, and Chinese Alliance for Helicobacter pylori Study. Chinese Consensus Report on Family-Based Helicobacter pylori Infection Control and Management (2021 Edition). Gut. 2022 Feb;71(2):238-253. doi: 10.1136/gutjnl-2021-325630. Epub 2021 Nov 26. PMID 34836916
- [Result] Lv ZF, Wang FC, Zheng HL, Wang B, Xie Y, Zhou XJ, Lv NH. Meta-analysis: is combination of tetracycline and amoxicillin suitable for Helicobacter pylori infection? World J Gastroenterol. 2015 Feb 28;21(8):2522-33. doi: 10.3748/wjg.v21.i8.2522. PMID 25741163
- [Result] Marko D, Calvet X, Ducons J, Guardiola J, Tito L, Bory F; GRESCA (Group for Eradication Studies from Catalonia and Aragon). Comparison of two management strategies for Helicobacter pylori treatment: clinical study and cost-effectiveness analysis. Helicobacter. 2005 Feb;10(1):22-32. doi: 10.1111/j.1523-5378.2005.00288.x. PMID 15691312
- [Result] Calvet X, Montserrat A, Guell M, Vergara M, Gene E. Ranitidine-bismuth citrate, tetracycline and metronidazole followed by triple therapy as alternative strategy for Helicobacter pylori treatment: a pilot study. Eur J Gastroenterol Hepatol. 2004 Oct;16(10):987-90. doi: 10.1097/00042737-200410000-00006. PMID 15371921
- [Result] Xie Y, Zhu Z, Wang J, Zhang L, Zhang Z, Lu H, Zeng Z, Chen S, Liu D, Lv N; the Chinese Study Group on Helicobacter pylori, Chinese Society of Gastroenterology. Ten-Day Quadruple Therapy Comprising Low-Dose Rabeprazole, Bismuth, Amoxicillin, and Tetracycline Is an Effective and Safe First-Line Treatment for Helicobacter pylori Infection in a Population with High Antibiotic Resistance: a Prospective, Multicenter, Randomized, Parallel-Controlled Clinical Trial in China. Antimicrob Agents Chemother. 2018 Aug 27;62(9):e00432-18. doi: 10.1128/AAC.00432-18. Print 2018 Sep. PMID 29914954
- [Result] Zhang J, Han C, Lu WQ, Wang N, Wu SR, Wang YX, Ma JP, Wang JH, Hao C, Yuan DH, Liu N, Shi YQ. A randomized, multicenter and noninferiority study of amoxicillin plus berberine vs tetracycline plus furazolidone in quadruple therapy for Helicobacter pylori rescue treatment. J Dig Dis. 2020 May;21(5):256-263. doi: 10.1111/1751-2980.12870. Epub 2020 Jun 9. PMID 32348007